CLINICAL TRIAL: NCT02290301
Title: An Observational Study to Evaluate Cardiovascular Outcomes of Patients With Type 2 Diabetes Mellitus Treated With Gemigliptin
Brief Title: An Observational Study to Evaluate Cardiovascular Outcomes of T2DM PatientsTreated With Gemigliptin
Status: Completed | Type: Observational
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-DPOS001
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LC15-0444

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus
  Interventions: Drug: gemigliptin

INTERVENTIONS:
Drug: gemigliptin

SUMMARY:
The primary objective of the study is to investigate cardiovascular safety of gemigliptin by evaluating the time until patients report with major adverse cardiovascular events (MACE) in T2DM patients treated with gemigliptin.

Study patients will be followed up to 4 years until MACE occurrence or until the patient drops out of the study or completion of the study. The patient who switches to a non-gemigliptin treatment after initiating gemigliptin therapy will be followed until MACE occurrence or until the patient drops out of the study or completion of the study.

The secondary objectives of the study are to evaluate adverse events related as well as not-related to MACE in diabetic patients treated with gemigliptin.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients, who are ≥ 19 years, with diagnosis of T2DM
* Diabetic patients whose condition cannot be adequately controlled by on-going dietary and/or under antidibatetic treatment are decided to prescribe gemigliptin according to the physician's judgment
* Patients must be willing and able to provide written informed consent form to use of personal information as well as the guardian's contact information and the permission to contact with the guardian in case the patient cannot be contacted.

Exclusion Criteria:

* Patients with T1DM
* Patients who experienced an acute coronary syndrome (ST-elevation myocardial infarction and non- ST elevation myocardial infarction) or ischemic stroke within the last 3 months before enrolment OR patients who have been treated with dipeptidyl peptidase IV (DPP-4) inhibitors or glucagon-like peptide (GLP-1) analogues for 3 months before enrolment.
* Patients with a diagnosis of severe or end-stage heart failure (New York Heart Association class III or IV).
* Patients who are currently participating or plan to participate in any interventional clinical trial
* Patients who are not prescribed gemigliptin or with counterindications for gemigliptin
* Patients who are considered not fit for the study by physician

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 5,000 Korean patients whose diabetic condition requires gemigliptin in monotherapy or in combination with other antidiabetic treatment, according to the physician's judgment, will be enrolled.
Sampling Method: Probability Sample
Enrollment: 5180 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Time-to-event for the primary composite MACE(Major Adverse Cardiovascular Events) endpoint | during the study period (2~4 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Kim EH, Kim SS, Kim DJ, Choi YS, Lee CW, Ku BJ, Cha KS, Song KH, Kim DK, Kim IJ. A prospective cohort study on effects of gemigliptin on cardiovascular outcomes in patients with type 2 diabetes (OPTIMUS study). Sci Rep. 2020 Nov 4;10(1):19033. doi: 10.1038/s41598-020-75594-5. PMID 33149182